CLINICAL TRIAL: NCT03302650
Title: Angiotensin II for Septic Shock Treatment: Effects On Macro- and Microcirculation A Randomized, Controlled Pilot Trial (ANGSTROM Trial)
Brief Title: Angiotensin II for Septic Shock Treatment
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The drug is not available
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-68-2017
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Angiotensin II; Saline Solution; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiotensin group (Experimental): Patients will receive Angiotensin II at a starting dose of 20 ng/Kg/min. During the first 30 minutes after randomization, the angiotensin II infusion will be titrated to achieve a mean arterial pressure of 65-75 mmHg while the norepinephrine infusion will be withdrawn and stopped. Following a stabilization of 60 minutes, the angiotensin II infusion is titrated to achieve a mean arterial pressure of 85-95 mmHg. Following a 30 minutes wash-in period and a 60 minutes stabilization period, a third set of measurements will be taken. Then, the angiotensin II infusion will be withdrawn in small steps and replaced by a norepinephrine infusion which will then be titrated to achieve a mean arterial pressure of 65-75 mmHg. Then, the final set of measurements will be taken.
  Interventions: Drug: Angiotensin II; Drug: Norepinephrine
- Normal saline group (Placebo Comparator): Patients will receive normal saline infusion in addition to norepinephrine infusion. The same mean arterial pressure levels (65-75 mmHg > 85-95 mmHg > 65-75 mmHg) will be achieved by titration of the norepinephrine infusion. Identical wash-in and stabilization periods will be kept as in the study group. Measurements will be taken at the same time points as in the study group. The maximum dose of norepinephrine applied will be 0.7 mcg/kg/min.
  Interventions: Drug: Normal saline; Drug: Norepinephrine

INTERVENTIONS:
Drug: Angiotensin II — Patients will receive angiotensin-II at a starting dose of 20 ng/Kg/min.
  Arms: Angiotensin group
Drug: Normal saline — Patients will receive normal saline.
  Arms: Normal saline group
Drug: Norepinephrine — patients will receive norepinephrine infusion adjusted according to blood pressure
  Other Names: Noradrenaline

SUMMARY:
This study aims to investigate the effect of angiotensin II on microcirculation and peripheral perfusion in patients with septic shock.

DETAILED DESCRIPTION:
Shock is a syndrome characterized by acute circulatory failure resulting in impaired peripheral tissue perfusion. Distributive shock is the most common type of shock and is usually caused by severe sepsis. Distributive shock is characterized by profound vasodilatation leading to decreased arterial blood pressure and impaired organ perfusion despite high cardiac output.

The use of vasopressors is an essential management line for distributive sock. Two groups of vasopressors are usually used for management of shock: catecholamines and vasopressin-like peptides. There is a continuous need for other vasopressors because:

1- Available vasopressors have narrow therapeutic window. 2- Patients with severe hypotension refractory to the currently available classes usually die.

A third system is usually engaged in the physiology of shock which is Renin-Angiotensin-aldosterone system. Angiotensin II is a natural hormone which is a potent vasopressor; moreover, angiotensin II stimulates the production of both antidiuretic hormone and adrenocorticotropin hormone.

In a pilot study, angiotensin II was reported as an effective rescue vasopressor in septic shock patients on multiple vasopressors. Angiotensin II improved mean arterial pressure and helped in reduction of the doses of catecholamines. In a recent large randomized controlled trial, angiotensin II improved blood pressure in catecholamine-resistant distributive shock patients.

Microcirculation is the primary site of oxygen and nutrient exchange. Maintenance of microcirculatory perfusion is a prerequisite for preservation of organ function. Multiple organ failure is common in patients with distributive shock despite maintenance of parameters of global perfusion due to disrupted microcirculatory perfusion. Furthermore, restoration of microcirculatory perfusion was correlated with improvement in survival. This study aims to investigate the effect of angiotensin II on peripheral microcirculation in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients.
* Aged above 18 years.
* With cardiac index > 2.4 L/min/BSA 1.73 m2.
* On high dose vasopressors (defined as norepinephrine infusion above 0.1 mcg/Kg/min)

Exclusion Criteria:

* Acute coronary syndrome.
* Impaired cardiac contractility
* Bronchospasm.
* Major burns
* Liver failure.
* Active bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Mean flow index | 6 Hours
  Mean flow index measured by Side stream dark field imaging optical probe (Microscan; MicroVision Medical, Amsterdam, Netherlands). Briefly, after gentle cleansing of the tongue by isotonic-saline-drenched gauze, avoiding pressure artifacts, 5 steady images of at least 20 seconds each will be obtained and stored under a random number. Offline blind analysis of each video will be done using a dedicated software (Automated Vascular Analysis 3.0; Academic Medical Center, University of Amsterdam, The Netherlands).
  The microvascular flow index (MFI) will be used to quantify microvascular blood flow. In this score, flow is characterized as absent (0), intermittent (1), sluggish (2), or normal (3), for each patient the values from 5 videos will be averaged. Since our investigation will be focused on small vessels, calculations will be separately performed for vessels with a diameter less than 20 ųm.

SECONDARY OUTCOMES:
Proportion of perfused vessels | 6 Hours
  Proportion of perfused vessels measured by Side stream dark field imaging optical probe (Microscan; MicroVision Medical, Amsterdam, Netherlands). Briefly, after gentle cleansing of the tongue by isotonic-saline-drenched gauze, avoiding pressure artifacts, 5 steady images of at least 20 seconds each will be obtained and stored under a random number. Offline blind analysis of each video will be done using a dedicated software (Automated Vascular Analysis 3.0; Academic Medical Center, University of Amsterdam, The Netherlands)
Perfused vessel density | 6 Hours
  Perfused vessel density measured by Side stream dark field imaging optical probe (Microscan; MicroVision Medical, Amsterdam, Netherlands). Briefly, after gentle cleansing of the tongue by isotonic-saline-drenched gauze, avoiding pressure artifacts, 5 steady images of at least 20 seconds each will be obtained and stored under a random number. Offline blind analysis of each video will be done using a dedicated software (Automated Vascular Analysis 3.0; Academic Medical Center, University of Amsterdam, The Netherlands)
systolic blood pressure | 6 hours
  systolic blood pressure measured in mmHg
Diastolic blood pressure | 6 hours
  diastolic blood pressure measured in mmHg
Heart rate | 6 hours
  heart rate in beats per minute
Serum lactate | 6 hours
  Serum lactate measured in milligrams per deciliter
Urine output | 6 hours
  quantity of urine in milliliters
Serum Creatinine | 24 hours
  serum creatinine measured in milligrams per deciliter
Serum Sodium | 24 hours
  Serum sodium measured in milligrams per deciliter
Serum potassium | 24 hours
  Serum potassium measured in milligrams per deciliter
Cardiac output | 6 hours
  quantity of blood pumper by the heart measured by electrical cardiometry in liters per minute
systemic vascular resistance | 6 hours
  systemic vascular resistance measured by electrical cardiometry
Norepinephrine requirements | 6 hours
  total requirement of norepinephrine needed to maintain mean arterial blood pressure above 65 mmHg
perfusion index | 6 hours
  proportion of pulsatile to non-pulsatile portions in peripheral circulation
total fluid intake | 24 hours
  amount of fluids received by the patient in milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department; Martin W Dünser, Professor, Study Director — Department of critical care, University of London college hospital
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided